CLINICAL TRIAL: NCT06688890
Title: Optimization of the Effectiveness of the Hydroalcoholic Solution of 3% Chlorhexidine Digluconate and 0.3% Potassium Sorbate in 70% Ethanol, Sorbectol, in Surgical Hand Preparation According to the UNE-EN 12791 Standard
Brief Title: Optimization of Surgical Hand Preparation Using Sorbectol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, MARIA DEL MAR PARRA RODRIGUEZ, podiatry and researcher in Health Sciences, Universidad Complutense de Madrid
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SORBUCM_MP
Record Dates: First submitted 2024-07-28; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hand Washing
Keywords: Sorbectol; bacterial load; inmediate effect; prolongated effect

STUDY DESIGN:
Intervention Model Description: clinical trial, randomized, crossover.
Who Masked: Participant
Masking Description: Participants ignore which product is being used in each intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1. Surgical hand rub with the reference product; n-propanol 60%. (Experimental)
  Interventions: Other: Surgical hand rub with the reference product; n-propanol 60%.
- 2. Surgical hand rub with the product P1; Sorbectol for 1 min. (Experimental)
  Interventions: Other: Surgical hand rub with the product P1; Sorbectol for 1 min.
- 3. Surgical hand rub with the product P2;Sorbectol for 3 min. (Experimental)
  Interventions: Other: Surgical hand rub with the product P2; Sorbectol for 3 min.
- 4. Surgical hand rub with the product P3; Sorbectol for 5 min. (Experimental)
  Interventions: Other: Surgical hand rub with the product P3; Sorbectol for 5 min.

INTERVENTIONS:
Other: Surgical hand rub with the reference product; n-propanol 60%. — Propanol hand rub for 3 min. The applied volume of product is sufficient to keep the hand moist for a total time of 3 min, adding as many 3 ml portions as necessary according to EN 12791. According to the EN 1279, the role assigned to each hand (immediate or 3h effect) in the first run is swapped in the subsequent runs.
  Arms: 1. Surgical hand rub with the reference product; n-propanol 60%.
Other: Surgical hand rub with the product P1; Sorbectol for 1 min. — Sorbectol hand rub for 1 min. The applied volume of product is sufficient to keep the hand moist for a total time of 1 min, adding as many 3 ml portions as necessary according to EN 12791. According to the EN 1279, the role assigned to each hand (immediate or 3h effect) in the first run is swapped in the subsequent runs.
  Arms: 2. Surgical hand rub with the product P1; Sorbectol for 1 min.
Other: Surgical hand rub with the product P2; Sorbectol for 3 min. — Sorbectol hand rub for 3 min. The applied volume of product is sufficient to keep the hand moist for a total time of 3 min, adding as many 3 ml portions as necessary according to EN 12791. According to the EN 1279, the role assigned to each hand (immediate or 3h effect) in the first run is swapped in the subsequent runs.
  Arms: 3. Surgical hand rub with the product P2;Sorbectol for 3 min.
Other: Surgical hand rub with the product P3; Sorbectol for 5 min. — Sorbectol hand rub for 5 min. The applied volume of product is sufficient to keep the hand moist for a total time of 5 min, adding as many 3 ml portions as necessary according to EN 12791. According to the EN 1279, the role assigned to each hand (immediate or 3h effect) in the first run is swapped in the subsequent runs.
  Arms: 4. Surgical hand rub with the product P3; Sorbectol for 5 min.

SUMMARY:
Previous studies evaluated the efficacy of the hydroalcoholic solution of 3% digluconate of chlorhexidine, 0.3% potassium sorbate and 70% ethanol, "Sorbectol" (Spanish patent ES 2 784 275 B2) in the surgical hand preparation with positive results. This clinical trial is focused on optimising the effectiveness of Sorbectol in the surgical hand preparation by scaling the application times of the product from 1 to 5 minutes following the test procedure and the effectiveness criteria of the European norm EN-12791.

DETAILED DESCRIPTION:
This is a randomised clinical trial with a Latin-square crossover design, to test the effectiveness of the Sorbectol solution in surgical hand preparation, according to the EN 12791 standard, at application times of 1, 3 or 5 minutes. The test compares the bacterial load on the hands of at least 23 healthy volunteers immediately (immediate effect) and three hours after (3-hour effect) application of the test product with respect to the reference product, RP, of EN 12791 (n-propanol 60%).

Briefly: The bacterial load on hands before antisepsis (pre-values) is obtained after the preparatory handwash using a diluted soft soap. Next, surgical hand antisepsis protocols are performed. Enrolled participants are randomly divided into four groups of the same size to receive RP or Sorbectol for 1 min (P1), 3 min (P2) or 5 min (P3) in parallel in a first run. The test is repeated in a second, third and fourth run changing the antisepsis roles for each group. A washout period of at least 2 weeks between experimental runs allow for the reconstitution of skin microbiota. All participants complete the four antiseptic procedures at the end of the trial.

The RP group, rub their hands with n-propanol (60% v/v) for 3 min. The test product groups, rub their hands with Sorbectol for 1 or 3 or 5 min. In all cases applying as many 3 ml portions as necessary to keep the hands moist for the selected time. After antisepsis the bacterial load (post-values) is determined using a split-hands model. One hand to assess the bacterial load immediately after treatment (immediate post-values) and the other hand to assess the bacterial load 3 hours later, keeping the hand gloved in the meantime (3-h post-values).

ELIGIBILITY:
Inclusion Criteria:

* Participants with healthy skin in both hands and short fingernails.
* No use of antibacterial agents for at least three days before the intervention.
* Not received antibiotic treatment for at least ten days before the intervention.

Exclusion Criteria:

* Known systemic pathologies.
* Wearing hand jewelry on the hands.
* Allergy to any ingredient of which the solutions used in the clinical trial are composed.
* Cognitive and / or motor limitation that makes it impossible to carry out instructions for hand washing.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-12-18 (Estimated); Study Completion 2024-12-18 (Estimated)

PRIMARY OUTCOMES:
Immediate effect assessed immediately after surgical hand antisepsis | Immediate effect is a measure determined at the time point 1, within the first 10 minutes of disinfection assay. The specific duration is subject to variation based on the particular application protocol of P1, P2, P3 and RP.]
  It refers to the reduction in bacterial load (expressed as the decimal logarithm, Log, of colony-forming units per milliliter of sample, CFU/ml) achieved immediately after the application of surgical hand antisepsis in one of the hands.
  The immediate effect is calculated by using the expression Log CFU/ml of immediate pre-values minus Log CFU/ml of immediate post-values, where the immediate pre-values are the bacterial counts pre-existing on the selected hand for immediate effect before disinfection, at the time point 0, and the immediate post-values are the bacterial counts determined on the same hand after the application of the antiseptic, at the time point 1.This primary outcome measure is used to evaluate the non-inferiority criterium proposed by the EN 12791 for tested antiseptic protocols, P1, P2 and P3 vs. RP.
Effect assessed 3-hours after surgical hand antisepsis | The 3-hours effect is a measure determined at the time point 2 which is 3 hours after the immediate effect determination]
  It refers to the reduction in bacterial load (expressed as the decimal logarithm, Log, of colony-forming units per milliliter of sample, CFU/ml) achieved 3 hours after of the surgical hand antisepsis on the opposite hand used for immediate effect determination.
  The 3-hours effect is calculated by using the expression Log CFU/ml of 3-hours pre-values minus Log CFU/ml of 3-hours post-values, where the 3-hours pre-values are the bacterial count pre-existing on the selected hand for 3-hours effect determination before disinfection, at the time point 0, and the 3-hours post-values are the bacterial count determined on the same hand 3-hours after the application of the antiseptic, at the time point 2.This primary outcome measure is used to evaluate the non-inferiority and sustained effect criteria proposed by the EN 12791 for tested antiseptic protocols, P1, P2 and P3 vs. RP.

SECONDARY OUTCOMES:
Bacterial counts preexisting on the hands before surgical hand antisepsis. Pre-values. | Prevalues is a measure determined at the time point 0 which represent the beginning of the disinfection assay
  This refers to the bacterial counts (expressed as the decimal logarithm, Log, of colony-forming units per milliliter of sample, CFU/ml) preexisting on the hands before surgical hand antisepsis. Preexisting bacterial counts are determined on each hand, in parallel at the time point 0. The bacterial count determined on one hand is called the immediate pre-value, and the bacterial count determined on the other hand is called the 3-hour pre-value This secondary outcome measure is used to calculate the extension of the immediate and 3-hours effect primary outcome measures for tested antiseptic protocols, P1, P2, P3 and the RP.
Bacterial counts immediately after surgical hand antisepsis. Immediate post-values | Immediate post-value is a measure determined at the time point 1, within the first 10 minutes of disinfection assay. The specific duration is subject to variation based on the particular application protocol of P1, P2, P3 and RP.]
  It refers to the bacterial count (expressed as the decimal logarithm, Log, of colony-forming units per milliliter of sample, CFU/ml) determined immediately after surgical hand antisepsis. This bacterial count, called the immediate post-value, is determined on the selected hand for immediate effect, at time point 1.
  This secondary outcome measure is used to calculate the extension of the immediate effect primary outcome measure for tested antiseptic protocols, P1, P2, P3 and the RP.
Bacterial counts 3-hours after surgical hand antisepsis. 3-hours post-values | 3-hours post-value is a measure determined at the time point 2, which is 3 hours after the immediate post-value determination.
  This refers to the bacterial count (expressed as the decimal logarithm, Log, of colony-forming units per milliliter of sample, CFU/ml) determined 3-hours after surgical hand antisepsis. This bacterial count, called the 3-hours post-value, is determined on the selected hand for 3-hours effect, at time point 2.
  This secondary outcome measure is used to calculate the extension of the 3-hours effect primary outcome measure for tested antiseptic protocols, P1, P2, P3 and the RP.

CONTACTS AND LOCATIONS:
Overall Officials: PARRA, Principal Investigator — UNIVERSIDAD COMPLUTENSE MADRID
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

REFERENCES:
- [Background] Rutala WA, Boyce JM, Weber DJ. Disinfection, sterilization and antisepsis: An overview. Am J Infect Control. 2023 Nov;51(11S):A3-A12. doi: 10.1016/j.ajic.2023.01.001. PMID 37890951
- [Background] Herraiz Soria E, Alou L, Martin-Villa C, Becerro-de-Bengoa-Vallejo R, Losa-Iglesias M, Sevillano D. Alcohol-Based Chlorhexidine and Potassium Sorbate Rub Strengthens the Effectiveness of Traditional Hand Scrubbing and Improves Long-Lasting Effectiveness-Evaluation of Hand Preparation Protocols According to EN 12791. Antibiotics (Basel). 2024 May 20;13(5):470. doi: 10.3390/antibiotics13050470. PMID 38786198